CLINICAL TRIAL: NCT00845845
Title: Fish Oil and Diet for the Treatment of Non-Alcoholic Steatohepatitis (NASH)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to low enrollment.
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Scott Cotler, MD, Professor of Medicine, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2003-0601
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Results first posted 2013-07-24 (Estimated); Last update posted 2013-07-24 (Estimated); Status verified 2013-06

CONDITIONS: Nonalcoholic Steatohepatitis (NASH); Hepatic Steatosis
Keywords: Non-alcoholic steatohepatitis; Omega-3 fatty acids; MRI; NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Fatty Liver | interventions — Omacor; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega-3-acid ethyl esters (Lovaza) (Active Comparator): Participants receive 4 milligrams (mg) daily of omega-3-acid ethyl esters (Lovaza) and dietary counseling for 24 weeks
  Interventions: Drug: Omega-3-acid ethyl esters (Lovaza)
- Placebo (Placebo Comparator): Participants receive daily placebo and dietary counseling for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Omega-3-acid ethyl esters (Lovaza) — 4 milligrams daily omega-3-acid ethyl esters (Lovaza) with dietary counseling for 24 weeks.
  Other Names: Lovaza
  Arms: Omega-3-acid ethyl esters (Lovaza)
Drug: Placebo — Daily placebo with dietary counseling for 24 weeks.
  Other Names: Sugar pill
  Arms: Placebo

SUMMARY:
The current pilot study assesses the use of magnetic resonance imaging (MRI) to quantify hepatic steatosis. It will provide preliminary data regarding the use of omega-3 fatty acid supplementation (Lovaza) for the treatment of nonalcoholic steatohepatitis (NASH).

ELIGIBILITY:
Inclusion Criteria:

* Males and females at least 18 years of age.
* Evidence of nonalcoholic steatohepatitis (NASH) on a liver biopsy performed within six months of entry to this study.
* Laboratory parameters indicative of decompensated liver disease including:

  * bilirubin less than 2 milligrams/decilitre (mg/dl).
  * stable albumin within normal limits.
  * prothrombin time less than 3 seconds prolonged.
* Serum creatinine less than 1.5 times the upper limit of normal.
* Diabetic patients must be stable on oral medication for diabetes or have had less than a 10 percent change in their insulin dose over the past two months.
* Thyroid stimulating hormone (TSH) or Free Thyroxine Index (FTI) within the normal range.
* Hepatitis C antibody negative.
* Hepatitis B Surface Antigen (HBsAg) seronegative.
* Antinuclear antibody (ANA) less than 1:320.
* Patient provides written informed consent.

Exclusion Criteria:

* Alcohol use exceeding 10 to 29 grams per day during the past six months.
* Evidence of a cause of liver disease other than nonalcoholic steatohepatitis (NASH) on liver biopsy including: viral hepatitis, alcoholic liver disease, autoimmune hepatitis, hemochromatosis, Wilson's disease, alpha-1 antitrypsin deficiency, or recent hepatoxic drug exposure.
* Patients with cirrhosis.
* Use of medications commonly associated with nonalcoholic steatohepatitis (NASH) including: glucocorticoids, estrogens, tamoxifen, methotrexate, nifedipine, diltiazem, chloroquine, isoniazid, or amiodarone within the past six months.
* Use of non-steroidal antiinflammatory drugs, fibrates (fenofibrate or gemfibrozil) or warfarin within one month of entering the study.
* Uncontrolled diabetes, defined as a glycated hemoglobin (A1C) level greater than 8%.
* Patients with insulin-dependent diabetes.
* History of jejunal-ileal bypass or extensive small bowel resection.
* Substance abuse including, but not limited to, alcohol or intravenous and inhaled drugs within the past six months.
* Use of chemotherapy within six months of enrollment.
* Patients taking metformin.
* Thyroid abnormality in which normal thyroid function cannot be maintained by medication.
* Pregnancy, females who are breastfeeding.
* Solid organ transplant recipient.
* History of a medical condition, which could interfere with participation in and completion of the protocol.
* Use of oral supplements of Vitamin E within one month of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-03; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Cotler, M.D., Principal Investigator — University of Illinois Chicago
Locations (1):
- The University of Illinois Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Reid AE. Nonalcoholic steatohepatitis. Gastroenterology. 2001 Sep;121(3):710-23. doi: 10.1053/gast.2001.27126. PMID 11522755
- [Background] Bacon BR, Farahvash MJ, Janney CG, Neuschwander-Tetri BA. Nonalcoholic steatohepatitis: an expanded clinical entity. Gastroenterology. 1994 Oct;107(4):1103-9. doi: 10.1016/0016-5085(94)90235-6. PMID 7523217
- [Background] Mofrad P, Contos MJ, Haque M, Sargeant C, Fisher RA, Luketic VA, Sterling RK, Shiffman ML, Stravitz RT, Sanyal AJ. Clinical and histologic spectrum of nonalcoholic fatty liver disease associated with normal ALT values. Hepatology. 2003 Jun;37(6):1286-92. doi: 10.1053/jhep.2003.50229. PMID 12774006
- [Background] Caldwell SH, Oelsner DH, Iezzoni JC, Hespenheide EE, Battle EH, Driscoll CJ. Cryptogenic cirrhosis: clinical characterization and risk factors for underlying disease. Hepatology. 1999 Mar;29(3):664-9. doi: 10.1002/hep.510290347. PMID 10051466
- [Background] Marrero JA, Fontana RJ, Su GL, Conjeevaram HS, Emick DM, Lok AS. NAFLD may be a common underlying liver disease in patients with hepatocellular carcinoma in the United States. Hepatology. 2002 Dec;36(6):1349-54. doi: 10.1053/jhep.2002.36939. PMID 12447858
- [Background] Neuschwander-Tetri BA, Caldwell SH. Nonalcoholic steatohepatitis: summary of an AASLD Single Topic Conference. Hepatology. 2003 May;37(5):1202-19. doi: 10.1053/jhep.2003.50193. PMID 12717402
- [Background] Chalasani N, Gorski JC, Asghar MS, Asghar A, Foresman B, Hall SD, Crabb DW. Hepatic cytochrome P450 2E1 activity in nondiabetic patients with nonalcoholic steatohepatitis. Hepatology. 2003 Mar;37(3):544-50. doi: 10.1053/jhep.2003.50095. PMID 12601351
- [Background] Li Z, Yang S, Lin H, Huang J, Watkins PA, Moser AB, Desimone C, Song XY, Diehl AM. Probiotics and antibodies to TNF inhibit inflammatory activity and improve nonalcoholic fatty liver disease. Hepatology. 2003 Feb;37(2):343-50. doi: 10.1053/jhep.2003.50048. PMID 12540784
- [Background] Listenberger LL, Han X, Lewis SE, Cases S, Farese RV Jr, Ory DS, Schaffer JE. Triglyceride accumulation protects against fatty acid-induced lipotoxicity. Proc Natl Acad Sci U S A. 2003 Mar 18;100(6):3077-82. doi: 10.1073/pnas.0630588100. Epub 2003 Mar 10. PMID 12629214
- [Background] Saxena NK, Ikeda K, Rockey DC, Friedman SL, Anania FA. Leptin in hepatic fibrosis: evidence for increased collagen production in stellate cells and lean littermates of ob/ob mice. Hepatology. 2002 Apr;35(4):762-71. doi: 10.1053/jhep.2002.32029. PMID 11915021
- [Background] Lavine JE. Vitamin E treatment of nonalcoholic steatohepatitis in children: a pilot study. J Pediatr. 2000 Jun;136(6):734-8. PMID 10839868
- [Background] Neuschwander-Tetri BA, Brunt EM, Wehmeier KR, Sponseller CA, Hampton K, Bacon BR. Interim results of a pilot study demonstrating the early effects of the PPAR-gamma ligand rosiglitazone on insulin sensitivity, aminotransferases, hepatic steatosis and body weight in patients with non-alcoholic steatohepatitis. J Hepatol. 2003 Apr;38(4):434-40. doi: 10.1016/s0168-8278(03)00027-8. PMID 12663234
- [Background] Marchesini G, Brizi M, Bianchi G, Tomassetti S, Zoli M, Melchionda N. Metformin in non-alcoholic steatohepatitis. Lancet. 2001 Sep 15;358(9285):893-4. doi: 10.1016/s0140-6736(01)06042-1. PMID 11567710
- [Background] Kudo N, Kawashima Y. Fish oil-feeding prevents perfluorooctanoic acid-induced fatty liver in mice. Toxicol Appl Pharmacol. 1997 Aug;145(2):285-93. doi: 10.1006/taap.1997.8186. PMID 9266801
- [Background] Neschen S, Moore I, Regittnig W, Yu CL, Wang Y, Pypaert M, Petersen KF, Shulman GI. Contrasting effects of fish oil and safflower oil on hepatic peroxisomal and tissue lipid content. Am J Physiol Endocrinol Metab. 2002 Feb;282(2):E395-401. doi: 10.1152/ajpendo.00414.2001. PMID 11788372
- [Background] Kris-Etherton PM, Harris WS, Appel LJ; Nutrition Committee. Fish consumption, fish oil, omega-3 fatty acids, and cardiovascular disease. Arterioscler Thromb Vasc Biol. 2003 Feb 1;23(2):e20-30. doi: 10.1161/01.atv.0000038493.65177.94. No abstract available. PMID 12588785
- [Background] Saito M, Kubo K. Relationship between tissue lipid peroxidation and peroxidizability index after alpha-linolenic, eicosapentaenoic, or docosahexaenoic acid intake in rats. Br J Nutr. 2003 Jan;89(1):19-28. doi: 10.1079/BJN2002731. PMID 12568661
- [Background] Meagher EA, Barry OP, Burke A, Lucey MR, Lawson JA, Rokach J, FitzGerald GA. Alcohol-induced generation of lipid peroxidation products in humans. J Clin Invest. 1999 Sep;104(6):805-13. doi: 10.1172/JCI5584. PMID 10491416
- [Background] Saad MF, Anderson RL, Laws A, Watanabe RM, Kades WW, Chen YD, Sands RE, Pei D, Savage PJ, Bergman RN. A comparison between the minimal model and the glucose clamp in the assessment of insulin sensitivity across the spectrum of glucose tolerance. Insulin Resistance Atherosclerosis Study. Diabetes. 1994 Sep;43(9):1114-21. doi: 10.2337/diab.43.9.1114. PMID 8070611
- [Background] Brunt EM, Janney CG, Di Bisceglie AM, Neuschwander-Tetri BA, Bacon BR. Nonalcoholic steatohepatitis: a proposal for grading and staging the histological lesions. Am J Gastroenterol. 1999 Sep;94(9):2467-74. doi: 10.1111/j.1572-0241.1999.01377.x. PMID 10484010

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twelve (12) individuals consented and were screened and nine (9) were randomized between March 2006 and June 2009. Due to low enrollment, the study was terminated in October 2010. Participants were recruited by study staff at outpatient clinics at The University of Illinois Chicago Hospitals and Clinics (UIHC).
Pre-assignment Details: A screening evaluation was used prior to group assignment to evaluate whether patients were affected by nonalcoholic steatohepatitis (NASH) and to evaluate the inclusion and exclusion criteria.
Period: Overall Study
Arm/Group | Omega-3-acid Ethyl Esters (Lovaza) | Placebo
Started | 3 | 6
Completed | 3 | 2
Not Completed | 0 | 4
Not completed — Lost to Follow-up | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Omega-3-acid Ethyl Esters (Lovaza) | Placebo | Total
Number analyzed (Participants) | 3 | 6 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 6 | 9
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 1 | 4 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 3
  Not Hispanic or Latino | 2 | 4 | 6
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Omega-3 Fatty Acid Supplementation and Its Effect on Hepatic Steatosis and Other Factors Associated With the Development of Nonalcoholic Steatohepatitis (NASH)
Time Frame: 24 weeks
Population: This study was terminated on October 12, 2010 due to low enrollment. Primary analyses were never completed.
Arm/Group | Omega-3-acid Ethyl Esters (Lovaza) | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Magnetic Resonance Imaging (MRI) as an Assessment of Hepatic Steatosis in Patients With Biopsy-proven Nonalcoholic Steatohepatitis (NASH)
Time Frame: 24 weeks
Population: This study was terminated on October 12, 2010 due to low enrollment. Primary analyses were never completed.
Arm/Group | Omega-3-acid Ethyl Esters (Lovaza) | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were captured using a systematic assessment from baseline (week 0) through week 24 for both the treatment and placebo groups.
Arm/Group | Omega-3-acid Ethyl Esters (Lovaza) | Placebo
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/6
Other Adverse Events (participants affected / at risk) | 2/3 | 0/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omega-3-acid Ethyl Esters (Lovaza) (N=3) | Placebo (N=6)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) — Herpes zoster is also known as shingles.
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omega-3-acid Ethyl Esters (Lovaza) (N=3) | Placebo (N=6)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated on October 12, 2010 due to low enrollment. Consequently, no analyses were completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes